CLINICAL TRIAL: NCT01945853
Title: Imaging Myelin Injury in Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Magnetic Resonance Imaging (MRI) in Amyotrophic Lateral Sclerosis (ALS)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Dr. Jeffrey Rothstein, Professor of Neurology, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NA_00080565
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 7 Tesla MRI (Experimental): 7T MRI will be done on ALS patients at baseline and at 6 month intervals.
  Interventions: Device: 7 Tesla MRI

INTERVENTIONS:
Device: 7 Tesla MRI

SUMMARY:
This is a pilot study to identify the degree of grey and white matter involvement in patients with Amyotrophic Lateral Sclerosis (ALS) utilizing non-invasive techniques. The imaging to be utilized will be the 7 Tesla (7T) magnetic resonance imaging (MRI) of the brain. These results will be correlated to the ALS Functional Rating Scale - Revised (ALSFRS-R) score to assess if any changes in MRI can be predictive in the disability of the ALS patients at baseline and at 6 month intervals. The participants will be asked to return every 6 months for a neurological examination, ALSFRS-R assessment, measurement of the vital capacity and MRI as outlined above to monitor progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females who are 18 - 80 years old.
* The participants will meet the standard diagnostic criteria for possible or probable ALS (based on El Escorial criteria). They will have been diagnosed by a Johns Hopkins Neurologist.
* Healthy controls will be recruited by their interest in assisting the ALS population.

Exclusion Criteria:

* Forced vital capacity less than 60 % of predicted value.
* Documented orthopnea on ALSFRS-R or otherwise unable to lie flat in an MRI scanner for the duration of the study.
* Presence of pacemakers, aneurysm clips, shrapnel or otherwise disallowed implanted metallic devices for obtaining an MRI scan.
* Pregnant or lactating females
* Glomerular filtration rate (GFR) less than 60
* History of: encephalitis, extensive white matter disease, intracranial hemorrhage, cerebral palsy, allergy to dye and/or IV drug abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
MRI Changes in ALS Patients Vs Healthy Controls | 2 years
  Voxel Based Morphometry will be utilized to look for any changes in the MRI results comparing ALS subjects to healthy volunteers.

SECONDARY OUTCOMES:
MRI Changes in ALS Patients | 2 years
  Voxel Based Morphometry will be utilized to look for any changes in the MRI results comparing ALS subjects comparing ALS subjects of differing clinical severity

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Rothstein, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States